CLINICAL TRIAL: NCT00402597
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Dose-Escalation and Dose-Confirmation Study to Evaluate the Safety and Efficacy of Rivaroxaban in Combination With Aspirin Alone or With Aspirin and a Thienopyridine in Subjects With Acute Coronary Syndromes
Brief Title: Rivaroxaban in Combination With Aspirin Alone or With Aspirin and a Thienopyridine in Patients With Acute Coronary Syndromes (The ATLAS ACS TIMI 46 Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Bayer (Industry)
Responsible Party: VP FRANCHISE MED LDR, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR013417; 39039039ACS2001; NCT01151332 (obsolete NCT alias)
Record Dates: First submitted 2006-11-21; First posted 2006-11-22 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome (ACS); Myocardial Ischemia; Rivaroxaban (BAY59-7939); Anti-platelet agents; Aspirin; Thienopyridine; Clopidogrel
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Ischemia | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 001 (Experimental): Rivaroxaban 1 rivaroxaban tablet twice daily for 6 months. Safety at each dose level will be confirmed before additional patients are randomized to the next higher dose level.
  Interventions: Drug: Rivaroxaban
- 002 (Experimental): Rivaroxaban/Placebo 1 rivaroxaban tablet once daily (and 1 placebo tablet once daily) for 6 months. Safety at each dose level will be confirmed before additional patients are randomized to the next higher dose level.
  Interventions: Drug: Rivaroxaban/Placebo
- 003 (Placebo Comparator): Placebo 1 placebo tablet twice daily for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivaroxaban/Placebo — 1 rivaroxaban tablet once daily (and 1 placebo tablet once daily) for 6 months. Safety at each dose level will be confirmed before additional patients are randomized to the next higher dose level.
  Arms: 002
Drug: Placebo — 1 placebo tablet twice daily for 6 months.
  Arms: 003
Drug: Rivaroxaban — 1 rivaroxaban tablet twice daily for 6 months. Safety at each dose level will be confirmed before additional patients are randomized to the next higher dose level.
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the safety of rivaroxaban in patients with recent acute coronary syndrome (ACS) and to assess the ability of rivaroxaban to reduce the occurrence of death, myocardial infarction (heart attack), repeat myocardial infarctions, stroke, and ischemia (inadequate blood supply to a local area) in patients with recent ACS.

DETAILED DESCRIPTION:
This is a randomized (patients will be assigned to study treatment by chance), double-blind (neither the patient nor the study doctor will know the identity of the assigned study treatment) study to evaluate the safety and efficacy of rivaroxaban (study drug) compared to placebo (a tablet identical in appearance to study drug but contains no active drug) in patients with acute coronary syndrome (ACS [a condition where blood flow in a blood vessel in the heart is restricted because of a blood clot]). Rivaroxaban is a drug that acts as a blood thinner and is being tested to see if it will be safe and effective in patients diagnosed ACS. The goal of this study is to identify the dose and dosing schedule (once-a-day or twice-a-day dosing) of rivaroxaban that will be safe and effective in preventing adverse cardiovascular outcomes such as death, myocardial infarctions (MI) including repeat myocardial infarction (reMI), stroke, or ischemia (inadequate blood supply to a local area) requiring revascularization (ie, the re-establishment of blood supply to a part or an organ) in patients with ACS who are receiving antiplatelet therapy (ie, aspirin alone or aspirin plus an approved thienopyridine, a type of drug such as clopidogrel that acts to inhibit the formation of blood clots). Approximately 3500 patients are planned to participate in the study for approximately 7 months. At study entry, all patients who are currently receiving treatment for ACS with antiplatelet therapy will be permitted to continue this therapy during the study. Patients will be enrolled and randomized to receive placebo, rivaroxaban administered as a once-daily dose, or rivaroxaban administered as a twice-daily dose at each dose level of rivaroxaban tested. Patients randomized at each dose level will continue to receive the same treatment for 6 months. Near the end of enrollment at the first dose level, available safety and efficacy data from patients will be assessed by an Operations Committee before enrolling and randomizing additional patients to the next higher dose level of rivaroxaban. Increasing dose levels of rivaroxaban are planned; however, progression to each higher dose level will be at the discretion of the Operations Committee. Patient safety will be monitored by evaluating adverse events reported, results from clinical laboratory tests, findings from electrocardiograms (ECGs) and vital signs measurements, findings from physical examinations, and the number of patients with protocol-defined major or minor bleeding, or bleeding requiring medical attention. All patients will take study drug or placebo tablets orally (by mouth) twice daily for 6 months starting at an initial total daily dose of 5 mg. Both once- and twice-daily dosing regimens will be tested at each rivaroxaban dose level planned.

ELIGIBILITY:
Inclusion Criteria:

* Have symptoms suggestive of ACS that lasted at least 10 minutes at rest occurring within 7 days of randomization
* Have a diagnosis of ST-elevation myocardial infarction or non-ST elevation myocardial infarction/unstable angina (ie, chest pain or discomfort) (ST elevation is an abnormal finding from an ECG test) with at least 1 protocol-defined high risk feature

Exclusion Criteria:

* Active bleeding or high risk of bleeding or intracranial hemorrhage (bleeding within the skull enclosing the brain)
* Need for continued anticoagulant therapy
* Significantly impaired renal (kidney) or hepatic (liver) function
* Severe concomitant diseases such as cardiogenic shock (heart damage that results in insufficient blood supply to other parts or organs of the body), refractory ventricular arrhythmias (irregular contractions of the heart unresponsive to treatment), or any severe condition that would limit life expectancy of the patient to less than 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3490 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Mega JL, Braunwald E, Mohanavelu S, Burton P, Poulter R, Misselwitz F, Hricak V, Barnathan ES, Bordes P, Witkowski A, Markov V, Oppenheimer L, Gibson CM; ATLAS ACS-TIMI 46 study group. Rivaroxaban versus placebo in patients with acute coronary syndromes (ATLAS ACS-TIMI 46): a randomised, double-blind, phase II trial. Lancet. 2009 Jul 4;374(9683):29-38. doi: 10.1016/S0140-6736(09)60738-8. Epub 2009 Jun 17. PMID 19539361
- [Derived] Gibson WJ, Nafee T, Travis R, Yee M, Kerneis M, Ohman M, Gibson CM. Machine learning versus traditional risk stratification methods in acute coronary syndrome: a pooled randomized clinical trial analysis. J Thromb Thrombolysis. 2020 Jan;49(1):1-9. doi: 10.1007/s11239-019-01940-8. PMID 31535314
- [Derived] Gibson CM, Mega JL, Burton P, Goto S, Verheugt F, Bode C, Plotnikov A, Sun X, Cook-Bruns N, Braunwald E. Rationale and design of the Anti-Xa therapy to lower cardiovascular events in addition to standard therapy in subjects with acute coronary syndrome-thrombolysis in myocardial infarction 51 (ATLAS-ACS 2 TIMI 51) trial: a randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of rivaroxaban in subjects with acute coronary syndrome. Am Heart J. 2011 May;161(5):815-821.e6. doi: 10.1016/j.ahj.2011.01.026. PMID 21570509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NCT00402597: Study 39039039ACS2001 (ATLAS ACS TIMI 46 Trial) was conducted at 297 centers in 27 countries between 17 November 2006 and 19 September 2008. A total of 3576 patients were screened for study and 3491 patients were randomly assigned to treatment.
Pre-assignment Details: Of the 3576 patients screened for study, 85 patients were screening failures and 3491 patients were randomly assigned to treatment. All randomized patients were included in the intent-to-treat (ITT) analysis set and were eligible for efficacy analyses. Of the 3491 patients, 29 never took study drug, leaving 3462 patients valid for safety analysis.
Groups:
- Placebo: One placebo tablet twice daily for 6 months.
- Riva 5 mg Total Daily Dose (TDD): Rivaroxaban 5 mg (2.5 mg twice a day or 5 mg once daily)
- Riva 10 mg TDD: Rivaroxaban 10 mg (5 mg twice a day or 10 mg once daily) for 6 months.
- Riva 15 mg TDD: Rivaroxaban 15 mg (7.5 mg twice a day or 15 mg once daily) for 6 months.
- Riva 20 mg TDD: Rivaroxaban 20 mg (10 mg twice a day or 20 mg once daily) for 6 months.
Period: Overall Study
Arm/Group | Placebo | Riva 5 mg Total Daily Dose (TDD) | Riva 10 mg TDD | Riva 15 mg TDD | Riva 20 mg TDD
Started | 1153 | 307 | 1046 | 353 | 603
Completed | 962 | 261 | 834 | 279 | 479
Not Completed | 191 | 46 | 212 | 74 | 124
Not completed — Death | 15 | 7 | 6 | 4 | 6
Not completed — Adverse Event | 81 | 18 | 106 | 39 | 71
Not completed — Lost to Follow-up | 8 | 1 | 8 | 2 | 3
Not completed — Withdrawal by Subject | 57 | 16 | 65 | 15 | 24
Not completed — reason not specified | 30 | 4 | 27 | 14 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Riva 5 mg Total Daily Dose (TDD) | Riva 10 mg TDD | Riva 15 mg TDD | Riva 20 mg TDD | Total
Number analyzed (Participants) | 1153 | 307 | 1046 | 353 | 603 | 3462
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 847 | 218 | 786 | 283 | 458 | 2592
  >=65 years | 306 | 89 | 260 | 70 | 145 | 870
Age Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.58) | 58.1 (9.76) | 57.2 (9.71) | 56.4 (9.38) | 57.4 (9.06) | 57.4 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 78 | 228 | 67 | 143 | 788
  Male | 881 | 229 | 818 | 286 | 460 | 2674
Region of Enrollment [Number; unit: participants]
  Australia | 75 | 14 | 73 | 15 | 29 | 206
  Belgium | 19 | 3 | 34 | 9 | 12 | 77
  Brazil | 11 | 0 | 26 | 0 | 0 | 37
  Bulgaria | 78 | 47 | 85 | 7 | 41 | 258
  Canada | 34 | 2 | 28 | 7 | 17 | 88
  China | 2 | 0 | 2 | 0 | 0 | 4
  Czech Republic | 48 | 0 | 58 | 33 | 41 | 180
  Denmark | 18 | 16 | 14 | 7 | 9 | 64
  Finland | 3 | 0 | 7 | 0 | 6 | 16
  France | 16 | 1 | 21 | 5 | 6 | 49
  Germany | 31 | 3 | 35 | 11 | 12 | 92
  Hungary | 11 | 0 | 14 | 7 | 4 | 36
  Israel | 43 | 0 | 26 | 16 | 11 | 96
  Italy | 43 | 3 | 56 | 17 | 17 | 136
  Korea (South) | 17 | 0 | 9 | 10 | 11 | 47
  Netherlands | 28 | 0 | 39 | 9 | 11 | 87
  New Zealand | 57 | 22 | 37 | 8 | 24 | 148
  Norway | 8 | 3 | 5 | 0 | 5 | 21
  Poland | 174 | 4 | 109 | 86 | 124 | 497
  Russia | 136 | 90 | 105 | 17 | 82 | 430
  Slovakia | 49 | 1 | 32 | 13 | 21 | 116
  South Africa | 6 | 0 | 7 | 0 | 4 | 17
  Spain | 35 | 5 | 36 | 12 | 15 | 103
  Sweden | 13 | 2 | 17 | 6 | 9 | 47
  Ukraine | 57 | 21 | 37 | 11 | 33 | 159
  United Kingdom | 9 | 1 | 19 | 15 | 8 | 52
  United States | 132 | 69 | 115 | 32 | 51 | 399

OUTCOME MEASURES:

1. Primary Outcome: Thrombolysis in Myocardial Infarction (TIMI) Clinically Significant Bleeding Events (Primary Safety)
Description: The number of patients with a first occurrence of a TIMI clinically significant bleeding event that occurred from the time of randomization to the time of the last patient contact. TIMI clinically significant bleeding events included TIMI minor bleeding events, TIMI major bleeding events, or any bleeding that required medical attention.
Time Frame: Day 1 to Day 210
Population: The safety population consisted of all randomized patients who took at least 1 dose of study medication after randomization during the double-blind treatment period.
Measure: Number; unit: Patients
Groups:
- Riva 5 mg Total Daily Dose (TDD): Rivaroxaban 5 mg (2.5 mg twice a day or 5 mg once daily) for 6 months.
Arm/Group | Placebo | Riva 5 mg Total Daily Dose (TDD) | Riva 10 mg TDD | Riva 15 mg TDD | Riva 20 mg TDD
Number analyzed (Participants) | 1153 | 307 | 1046 | 353 | 603
Patients | 36 | 17 | 109 | 43 | 89

2. Primary Outcome: The Composite Endpoint of All Cause Death, Myocardial Infarction (MI) (Including Repeat MI), Stroke (Ischemic, Hemorrhagic or Unknown), or Severe Recurrent Ischemia Requiring Revascularization (Primary Efficacy)
Description: The number of patients who died due to any cause or had a first occurrence of MI (including repeat MI) or stroke (ischemic, hemorrhagic or unknown) or severe recurrent ischemia requiring revascularization from the time of randomization to the last date of patient contact.
Time Frame: Day 1 to Day 210
Population: The intent-to-treat (ITT) population consisted of all patients who were randomized to treatment, regardless of study drug intake.
Measure: Number; unit: Patients
Arm/Group | Placebo | Riva 5 mg Total Daily Dose (TDD) | Riva 10 mg TDD | Riva 15 mg TDD | Riva 20 mg TDD
Number analyzed (Participants) | 1160 | 308 | 1056 | 356 | 611
Patients | 83 | 23 | 55 | 27 | 36

3. Secondary Outcome: The Composite Endpoint of Death (All Cause), Myocardial Infarction (MI) (or Repeat MI), or Stroke
Description: The number of patients who died due to any cause or had a first occurrence of MI (or repeat MI) or stroke from the time of randomization to the last date of patient contact.
Time Frame: Day 1 to Day 210
Population: The ITT population consisted of all patients who were randomized to treatment, regardliess of study drug intake.
Measure: Number; unit: Patients
Arm/Group | Placebo | Riva 5 mg Total Daily Dose (TDD) | Riva 10 mg TDD | Riva 15 mg TDD | Riva 20 mg TDD
Number analyzed (Participants) | 1160 | 308 | 1056 | 356 | 611
Patients | 66 | 18 | 40 | 21 | 22

4. Secondary Outcome: The Composite Endpoint of Cardiovascular Death, Myocardial Infarction (MI), or Stroke
Description: The number of patients with the composite endpoint of cardiovascular death or MI or stroke that occurred from the time of randomization to the last date of patient contact.
Time Frame: Day 1 to Day 210
Population: The ITT population consisted of all patients who were randomized to treatment regardless of study drug intake.
Measure: Number; unit: Patients
Arm/Group | Placebo | Riva 5 mg Total Daily Dose (TDD) | Riva 10 mg TDD | Riva 15 mg TDD | Riva 20 mg TDD
Number analyzed (Participants) | 1160 | 308 | 1056 | 356 | 611
Patients | 63 | 18 | 40 | 21 | 21

5. Secondary Outcome: The Number of Deaths (All Cause)
Description: The number of patients who died due to any cause from the time of randomization to the last date of patient contact.
Time Frame: Day 1 to Day 210
Population: The ITT population consisted of all patients who were randomized to treatment, regardless of study drug intake.
Measure: Number; unit: Patients
Arm/Group | Placebo | Riva 5 mg Total Daily Dose (TDD) | Riva 10 mg TDD | Riva 15 mg TDD | Riva 20 mg TDD
Number analyzed (Participants) | 1160 | 308 | 1056 | 356 | 611
Patients | 18 | 11 | 9 | 4 | 9

6. Secondary Outcome: The Composite Endpoint of Death (All Cause), MI (or reMI), Stroke, Severe Recurrent Ischemia Requiring Revascularization, or Thrombolysis in Myocardial Infarction (TIMI) (Major or Minor Bleeding) to Assess the Net Clinical Benefit
Description: The number of patients who died due to any cause or had a first occurrence of MI (or repeat MI), or stroke, or severe recurrent ischemia requiring revascularization, or TIMI (major or minor bleeding) from the time of randomization to the last date of patient contact to assess the net clinical benefit of rivaroxaban.
Time Frame: Day 1 to Day 210
Population: The ITT population consisted of all patients who were randomized to treatment, regardless of study drug intake.
Measure: Number; unit: Patients
Arm/Group | Placebo | Riva 5 mg Total Daily Dose (TDD) | Riva 10 mg TDD | Riva 15 mg TDD | Riva 20 mg TDD
Number analyzed (Participants) | 1160 | 308 | 1056 | 356 | 611
Patients | 88 | 24 | 71 | 35 | 48

ADVERSE EVENTS:
Description: Only Treatment-Emergent Adverse Events are presented in the following sections, called as Frequent Adverse Events and Serious Adverse Events
Arm/Group | Placebo | Riva 5 mg Total Daily Dose (TDD) | Riva 10 mg TDD | Riva 15 mg TDD | Riva 20 mg TDD
Serious Adverse Events (participants affected / at risk) | 247/1153 | 74/307 | 208/1046 | 72/353 | 128/603
Other Adverse Events (participants affected / at risk) | 223/1153 | 67/307 | 293/1046 | 108/353 | 148/603
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1153) | Riva 5 mg Total Daily Dose (TDD) (N=307) | Riva 10 mg TDD (N=1046) | Riva 15 mg TDD (N=353) | Riva 20 mg TDD (N=603)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0 | 1
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 3 | 0 | 1 | 0 | 2
Acute Myocardial Infarction (Cardiac disorders) | 28 | 6 | 13 | 8 | 5
Angina Pectoris (Cardiac disorders) | 22 | 4 | 16 | 4 | 10
Angina Unstable (Cardiac disorders) | 42 | 12 | 23 | 11 | 21
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Arteriospasm Coronary (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 7 | 5 | 6 | 2 | 1
Atrial Flutter (Cardiac disorders) | 1 | 0 | 3 | 0 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 2 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 2 | 0 | 0 | 0 | 3
Cardiac Failure (Cardiac disorders) | 6 | 1 | 6 | 1 | 0
Cardiac Failure Acute (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 3 | 1 | 3 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiogenic Shock (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 5 | 0 | 3 | 1 | 0
Coronary Artery Insufficiency (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Coronary Artery Stenosis (Cardiac disorders) | 1 | 1 | 0 | 2 | 0
Dressler's Syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Intracardiac Thrombus (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Left Ventricular Failure (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 5 | 3 | 6 | 3 | 8
Myocardial Ischaemia (Cardiac disorders) | 6 | 1 | 12 | 1 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 3 | 1 | 0
Parasystole (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 2 | 0 | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Postinfarction Angina (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular Fibrillation (Cardiac disorders) | 1 | 0 | 1 | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1 | 2 | 0 | 1
Endocardial Fibroelastosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Thyroid Disorder (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Conjunctival Haemorrhage (Eye disorders) | 1 | 1 | 0 | 0 | 0
Eye Haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 1
Retinal Artery Thrombosis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vitreous Haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anal Fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 1 | 10 | 3 | 6
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gingival Bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophageal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Peptic Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Retroperitoneal Haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 3
Catheter Site Haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0
Chest Discomfort (General disorders) | 1 | 1 | 2 | 0 | 2
Chest Pain (General disorders) | 24 | 9 | 17 | 2 | 9
Death (General disorders) | 0 | 1 | 0 | 0 | 0
Injection Site Phlebitis (General disorders) | 0 | 1 | 0 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 11 | 4 | 13 | 2 | 5
Puncture Site Haemorrhage (General disorders) | 0 | 0 | 2 | 0 | 1
Puncture Site Reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 1
Sudden Cardiac Death (General disorders) | 3 | 1 | 1 | 0 | 1
Sudden Death (General disorders) | 0 | 0 | 2 | 1 | 0
Vessel Puncture Site Haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 1 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 1 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 2
Anaphylactic Shock (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Abscess Limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Anal Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 2
Cellulitis (Infections and infestations) | 2 | 1 | 1 | 0 | 1
Cellulitis Orbital (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis Pharyngeal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 2 | 0 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gingival Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Implant Site Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 1 | 3 | 0
Post Procedural Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Wound Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 2
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Implantable Defibrillator Malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 0 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Skull Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0 | 0
Thrombosis in Device (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 0 | 1
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 1 | 0
Vascular Pseudoaneurysm Ruptured (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 2 | 1 | 0 | 1
Angiogram (Investigations) | 0 | 0 | 0 | 1 | 0
Arteriogram Coronary (Investigations) | 6 | 0 | 3 | 1 | 4
Aspartate Aminotransferase Increased (Investigations) | 0 | 2 | 0 | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Bilirubin Increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 0 | 1 | 0 | 0
C-Reactive Protein Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Chest X-Ray Abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Ejection Fraction Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 1 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 1 | 0 | 0 | 0
Liver Function Test Abnormal (Investigations) | 2 | 0 | 0 | 0 | 0
Occult Blood (Investigations) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Arthritis Reactive (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Breast Cancer in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ovarian Granulosa-Theca Cell Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Brain Oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 2 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Motor Neurone Disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 2 | 0 | 0 | 0 | 1
Progressive Supranuclear Palsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 2 | 0 | 1
Vascular Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Acute Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Drug Dependence (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Major Depression (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Calculus Ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3
Renal Colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Renal Haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 2 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 3 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Angioplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Catheterisation Cardiac (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 1
Coronary Artery Bypass (Surgical and medical procedures) | 3 | 2 | 2 | 0 | 2
Coronary Revascularisation (Surgical and medical procedures) | 1 | 0 | 4 | 0 | 2
Elective Procedure (Surgical and medical procedures) | 2 | 0 | 1 | 0 | 0
Elective Surgery (Surgical and medical procedures) | 1 | 1 | 0 | 0 | 0
Implantable Defibrillator Insertion (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Percutaneous Coronary Intervention (Surgical and medical procedures) | 5 | 1 | 6 | 1 | 2
Surgery (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Aortic Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Aortic Stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Arteriovenous Fistula (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Femoral Arterial Stenosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Femoral Artery Occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 5 | 0 | 2
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Iliac Artery Occlusion (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Intermittent Claudication (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Neovascularisation (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1153) | Riva 5 mg Total Daily Dose (TDD) (N=307) | Riva 10 mg TDD (N=1046) | Riva 15 mg TDD (N=353) | Riva 20 mg TDD (N=603)
Angina Pectoris (Cardiac disorders) | 44 | 16 | 43 | 8 | 22
Gingival Bleeding (Gastrointestinal disorders) | 13 | 4 | 47 | 32 | 33
Chest Pain (General disorders) | 91 | 26 | 99 | 31 | 48
Contusion (Injury, poisoning and procedural complications) | 33 | 8 | 40 | 18 | 31
Dizziness (Nervous system disorders) | 47 | 16 | 32 | 9 | 18
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 | 11 | 89 | 44 | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less